CLINICAL TRIAL: NCT03171337
Title: To Explore the Cerebral Function Efficacy of Acupuncture and Fu's Subcutaneous Needling (FSN) in the Treatment of Chronic Tension-type Headache by Means of fMRI: a Single-blinded, Randomized Controlled Trials.
Brief Title: The Efficacy of Acupuncture and Fu's Subcutaneous Needling (FSN ) in Treating Chronic Tension-type Headache by fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiang Xumei (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Jiang Xumei, Postdoctor;Lecturer, South China Normal University
Organization: South China Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SouthSNU
Record Dates: First submitted 2017-05-04; First posted 2017-05-31 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Chronic Tension-Type Headache
Keywords: Chronic tension-type headache; Acupuncture; Fu's subcutaneous needling(FSN); fMRI; Regional homogeneity (ReHo)
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The parallel group includes the positive and negative controls, the positive control is Fu's Subcutaneous Needling group and the negative is Sham acupuncture group. And the other parallel control is the fMRI of patients with CTTH VS fMRI of healthy people.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupuncture (Experimental): Acupuncture at acupoints for CTTH according to TCM theory, twice 1 week for 4 weeks，fMRI will be used to detect the cerebral function changes
  Interventions: Device: Acupuncture
- Fu's subcutaneous needling (FSN) (Active Comparator): FSN at the points related with CTTH, twice 1 week for 4 weeks, fMRI will be used to detect the cerebral function changes.
  Interventions: Device: Fu's Subcutaneous Needling (FSN)
- Sham acupuncture (Sham Comparator): Streitberger placebo needles at nonacupoint for CTTH, twice 1 week for 4 weeks,fMRI will be used to detect the cerebral function changes.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture at acupoints for CTTH according to TCM theory using stainless filiform needle.
  Other Names: Filiform needle
  Arms: Acupuncture
Device: Fu's Subcutaneous Needling (FSN) — Fu's subcutaneous needling at specific points for CTTH using soft casing needle.
  Other Names: Fu's Acupuncture; Floating Needling; Fu Needling
  Arms: Fu's subcutaneous needling (FSN)
Device: Sham acupuncture — Sham acupuncture at non-acupoints using Steinberger placebo needles
  Other Names: Placebo Acupuncture
  Arms: Sham acupuncture

SUMMARY:
Epidemiological studies show a one-year prevalence of 30%-60% for episodic tension-type headache (TTH) and 2%-3% for chronic TTH (CTTH). Many TTH patients seek acupuncture treatment worldwide, and CTTH is one of the most commonly treated. FSN has been used to treat CTTH recently; the curative effect of it was especially good for CTTH accompanying pericranial tenderness. Nonetheless, the effectiveness of acupuncture and FSN for CTTH remains controversial. Several research results showed that symptoms of TTH improve after acupuncture treatment, but these improvements were more subjective than objective measures. So, the aim of this study is to determine the cerebral function efficacy of acupuncture and FSN in the treatment of CTTH, using Headache impact test questionnaire (HIT-6), VAS to evaluate the subjective symptom and fMRI to detect the objective cerebral function changes.

Intervention: device: acupuncture; Fu's subcutaneous; placebo sham acupuncture

DETAILED DESCRIPTION:
Tension-type headache (TTH) is the most prevalent type of primary headache. Unlike migraine, however, there have been no significant treatment advances for chronic TTH in the past few decades, probably due to the limited understanding of its pathophysiology compared with that of migraine. The objective of the present study is to investigate the cerebral function imaging changes in patients with chronic tension headache trough comparing that in healthy people, focus on the regional homogeneity (ReHo) of ROIs of brain. In addition, the effect of acupuncture and Fu's subcutaneous needing (FSN) on the cerebral function will also be studied. This is a clinical trial study, randomized, in parallel, single-blinded assessor, and with a sham placebo control.

The study will be carried out in the （Traditional therapy center, Guangdong Hospital of Traditional Chinese Medicine）. Patients will be collected according to the inclusion criteria (conform to diagnose criterion for headache ICHD-3), with age between 18 and 45 years old. Healthy people will be collected too according to the inclusion criteria for healthy people, with age matching with the patients. The participants will respond to questionnaires at the beginning and end of the first, fifth and last therapeutic intervention and their fMRI of brain will be acquired. The therapeutic intervention will include: 8 acupuncture sessions, 8 FSN sessions and 8 placebo sham acupuncture sessions (twice per week for 4 weeks). The measurements taken will be: impact of headache on daily life, severity of headache, emotional problem of headache, the cerebral function of ROIs (by means of fMRI) of headache and so on.

Through these interventions it is hoped that patients will present an improvement in their pain presentation, quality of life and emotional problem, as well as cerebral function imaging in certain region of brain. Evidence for these hypotheses will provide the cerebral function effect mechanism of acupuncture and FSN to CTTH, and some evidence in the research will perhaps support that acupuncture and FSN are two type minimally-invasive treatment methods, with few side-effects and low cost.

ELIGIBILITY:
Inclusion Criteria:

1. Conforms to clinical diagnostic criteria of CTTH associated with pericranial tenderness（ICHD-3 beta version）, Han nationality.
2. Aged between 18 and 45 years old men or women with right-handed.
3. No history of cognitive dysfunction.
4. Seeking medical advice for TTH for the first time.
5. Providing informed consent to participate in the study.

Exclusion Criteria:

1. Taking analgesics or other drugs may affect the resting state fMRI scans of brain within two weeks.
2. Have hypertension, diabetes, anxiety, depression and other systemic diseases, other chronic pain etc. Psychiatric or neurologic disorder that unable patient to consent and follow study protocol.
3. Combined with other type headache.
4. Intracranial lesions are found in MRI or CT scans.
5. Headache breaks out within 24h after fMRI scan.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-06-10 (Estimated); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Regional homogeneity data (ReHo) (using Kendall's coefficient of concordance as index) of Resting state fMRI of the whole brain (from the Vertex to Basicranial) | 5 months
  ReHo data before and after the first/last, as well as after the fourth acupuncture, FSN and sham acupuncture treatment, Changes of ReHo data from baseline to after the first, fourth, last treatment will be calculated in each treatment group and will be compared with each other.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS） | 4 months.
  The intensity of pain was measured by a 10 cm VAS. The scores range from no pain (zero) to the worst possible pain (10 cm).
Headache Impact Test (HIT-6) | 4 months.
  It consists of six questions that assess the impact of headache on the ability to work, study, at home and in social situations.

CONTACTS AND LOCATIONS:
Overall Officials: Zhouyi Guo, Pro, Study Chair — SATCM Third Grade Laboratory of Chinese Medicine and Photonics Technology, College of Biophotonics and fMRI chamber, research resources center, South China Normal University.; Jian Sun, PhD, Principal Investigator — Traditional therapy center, Guangdong Hospital of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided